CLINICAL TRIAL: NCT05219409
Title: Effects of Sitagliptin in Relatives of Patients With Type 1 Diabetes Mellitus, at High Risk of Developing the Disease
Brief Title: Effects of Sitagliptin in Relatives of T1D Patients
Acronym: SITA-one
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Paolo Fiorina, MD, Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 01/2022
Record Dates: First submitted 2022-01-20; First posted 2022-02-02 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Type 1 Diabetes
Keywords: Sitagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Intervention Model Description: A randomized controlled open label intervention study is proposed. Relatives of patients with type 1 diabetes in stage 2 will be included in the study and divided into two groups by randomization: sitagliptin add-on therapy vs placebo(group of control)
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment group (Active Comparator): Sitagliptin
  Interventions: Drug: Sitagliptin; Device: Professional CGM
- Control group (Placebo Comparator): Placebo
  Interventions: Device: Professional CGM

INTERVENTIONS:
Drug: Sitagliptin — The dose of sitagliptin will be established on the basis of the estimated glomerular filtrate: 100 mg in single daily administration (estimated glomerular filtration rate less than or equal to 45 mL / min / 1.73 m2) or 50 mg (estimated glomerular filtration rate 30-45 mL / min / 1.73 m2)
  Arms: Treatment group
Device: Professional CGM — The sensor records the patient's glucose readings every 15 minutes for up to 14 days.

SUMMARY:
Type 1 Diabetes (T1D) is a chronic autoimmune disease, with a genetic background, resulting from the immune-mediated destruction of beta cells of the pancreas. It can lead to fatal short-term and long-term complications, especially if it is diagnosed late. Three stages of the disease can be identified: Stage 1 is defined by the presence of two or more anti-islet autoantibodies (GAD65, ICA, IA-2, ZnT8) with normoglycemia, Stage 2 shows progression to dysglycemia (impaired glucose tolerance) in the setting of two or more anti-islet autoantibodies, Stage 3 occurs when a patient meets ADA criteria for the diagnosis of diabetes. It's been demonstrated that Teplizumab (an Fc receptor nonbinding anti-CD3 monoclonal antibody) delays the transition from pre-symptomatic T1D (stage 2) to overt T1D (stage 3). Also Sitagliptin, a DPP4 inhibitor, has been proved effective in inhibiting inflammation in T1D both in vitro in T1D mice, and in vivo in Latent autoimmune diabetes in adults (LADA) patients. Furthermore, it has been confirmed that Sitagliptin reduces the prevalence of worse forms of acute GVHD after myeloablative allogeneic hematopoietic stem-cell transplantation.

The study aims to investigate if Sitagliptin can have a delaying effect on progression to overt T1D, on the account of its anti-inflammatory properties. The cohort is made of screened relatives of T1D patients, who are classified as high-risk of developing T1D.

Screening relatives of T1D patients for dysglycemia and anti-islet autoantibodies. Selecting the patients in Stage 2 Pre-symptomatic T1D (dysglycemia and at least two types of autoantibodies) and then beginning therapy with Sitagliptin, while monitoring their glucose metabolism with a Continuous Glucose Monitoring (CGM) system.

ELIGIBILITY:
Inclusion Criteria:

* Age of the subject between 10 and 45 years
* Subject (or legal guardian in the case of a minor) is able to provide informed consent
* If a first degree relative of the proband with T1D must be between 6 and 45 years old (brother, sister, parent, child)
* If a relative of the proband with T1D is second degree, he must be between 6 and 20 years old (nephew, uncle, aunt, grandfather, grandmother, cousin)
* Presence of at least two autoantibodies associated with diabetes
* Impaired glucose tolerance on the OGTT test (fasting glucose greater than 110 mg/dl but less than 126 mg/dl or 2-hour glucose greater than or equal to 140 mg/dl but less than 200 mg/dl or 'OGTT at 30', 60 ', 90' greater than or equal to 200 mg/dl)
* If the subject is a female with reproductive potential, she must have a negative pregnancy test at the enrollment visit and must agree not to seek pregnancy for at least one year from randomization
* If the subject is male, he must agree not to seek pregnancies with any partner for at least one year from the randomization
* The subject must agree to renounce other types of trials during this study
* Weight at the time of recruitment of at least 26 kg
* It must be favorable and clinically acceptable to postpone vaccinations with live and attenuated agents for at least one year after treatment

Exclusion Criteria:

* Type 1 Diabetes Mellitus previously diagnosed or diagnosed during screening investigations
* Serological evidence of current or past HIV, Hepatitis C, Hepatitis B
* Changes in blood counts, INR or liver enzymes
* Being pregnant or breastfeeding
* Evidence of pancreatic changes in the laboratory
* Having undergone a previous experimental treatment for Type 1 Diabetes Mellitus
* Chronic Renal Failure stage IIIa onwards (eGFR <45 ml / min / 1.7 m2)
* History of previous pancreatitis
* Lymphopenia (<1000 lymphocytes / µL)
* Neutropenia (<1500 PMN / µL)
* Thrombocytopenia (<150,000 platelets / µL)
* Anemia (Hgb <10 grams / deciliter [g / dL])
* AST or ALT> 1.5 x ULN
* Total bilirubin> 1.5 x upper limit of normal (ULN) with the exception of subjects diagnosed with Gilbert's syndrome who may be eligible provided they have no other cause leading to hyperbilirubinemia
* INR> 0.1 above the upper limit of the norm at the laboratory of the participating center
* Alterations of Amylase and Lipase due to the pancreas
* Chronic active infection other than localized skin infections
* A positive PPD test
* Vaccination with a live virus within 8 weeks of randomization
* Vaccination with a killed virus within 4 weeks of randomization
* Laboratory or clinical evidence of acute EBV or CMV infection
* Serological evidence of current or past HIV, hepatitis B or hepatitis C infection
* Being currently pregnant or breastfeeding, or planning to become pregnant
* Chronic use of steroids or other immunosuppressive agents
* A history of asthma or atopic disease that requires chronic treatment
* Untreated hypothyroidism or active Graves' disease at randomization
* Current use of non-insulin drugs that affect glycemic control
* Previous OKT®3 or other anti-CD3 treatment
* Administration of a monoclonal antibody within the year prior to randomization
* Participation in any type of clinical trial of therapeutic drugs or vaccines in the 12 weeks prior to randomization
* Any conditions that, in the opinion of the investigator, could interfere with the conduct of the study or with the safety of the subject.

Ages: 10 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of new diagnoses of Type 1 Diabetes Mellitus per year | 3 years

SECONDARY OUTCOMES:
Number of participants with adverse effects on Sitagliptin | 3 years

OTHER OUTCOMES:
To study the effects of Sitagliptin on metabolic markers (C-peptide, OGTT, Insulin) over time up to the diagnosis of diabetes | 3 years
To study the prevalence of T1D, T1D-related Auto-antibodies and Dysglycemia in relatives of T1D patients | 3 years
Monitor Stage 2 patients with a CGM system (continuous blood glucose detection) | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- ASST FBF Sacco, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Variation and trends in incidence of childhood diabetes in Europe. EURODIAB ACE Study Group. Lancet. 2000 Mar 11;355(9207):873-6. PMID 10752702
- [Result] Eisenbarth GS. Type I diabetes mellitus. A chronic autoimmune disease. N Engl J Med. 1986 May 22;314(21):1360-8. doi: 10.1056/NEJM198605223142106. No abstract available. PMID 3517648
- [Result] Ziegler AG, Rewers M, Simell O, Simell T, Lempainen J, Steck A, Winkler C, Ilonen J, Veijola R, Knip M, Bonifacio E, Eisenbarth GS. Seroconversion to multiple islet autoantibodies and risk of progression to diabetes in children. JAMA. 2013 Jun 19;309(23):2473-9. doi: 10.1001/jama.2013.6285. PMID 23780460
- [Result] Dabelea D, Pihoker C, Talton JW, D'Agostino RB Jr, Fujimoto W, Klingensmith GJ, Lawrence JM, Linder B, Marcovina SM, Mayer-Davis EJ, Imperatore G, Dolan LM; SEARCH for Diabetes in Youth Study. Etiological approach to characterization of diabetes type: the SEARCH for Diabetes in Youth Study. Diabetes Care. 2011 Jul;34(7):1628-33. doi: 10.2337/dc10-2324. Epub 2011 Jun 2. PMID 21636800
- [Result] Insel RA, Dunne JL, Atkinson MA, Chiang JL, Dabelea D, Gottlieb PA, Greenbaum CJ, Herold KC, Krischer JP, Lernmark A, Ratner RE, Rewers MJ, Schatz DA, Skyler JS, Sosenko JM, Ziegler AG. Staging presymptomatic type 1 diabetes: a scientific statement of JDRF, the Endocrine Society, and the American Diabetes Association. Diabetes Care. 2015 Oct;38(10):1964-74. doi: 10.2337/dc15-1419. PMID 26404926
- [Result] Sosenko JM, Skyler JS, Mahon J, Krischer JP, Greenbaum CJ, Rafkin LE, Beam CA, Boulware DC, Matheson D, Cuthbertson D, Herold KC, Eisenbarth G, Palmer JP; Type 1 Diabetes TrialNet and Diabetes Prevention Trial-Type 1 Study Groups. Use of the Diabetes Prevention Trial-Type 1 Risk Score (DPTRS) for improving the accuracy of the risk classification of type 1 diabetes. Diabetes Care. 2014 Apr;37(4):979-84. doi: 10.2337/dc13-2359. Epub 2014 Feb 18. PMID 24550217
- [Result] Herold KC, Bundy BN, Long SA, Bluestone JA, DiMeglio LA, Dufort MJ, Gitelman SE, Gottlieb PA, Krischer JP, Linsley PS, Marks JB, Moore W, Moran A, Rodriguez H, Russell WE, Schatz D, Skyler JS, Tsalikian E, Wherrett DK, Ziegler AG, Greenbaum CJ; Type 1 Diabetes TrialNet Study Group. An Anti-CD3 Antibody, Teplizumab, in Relatives at Risk for Type 1 Diabetes. N Engl J Med. 2019 Aug 15;381(7):603-613. doi: 10.1056/NEJMoa1902226. Epub 2019 Jun 9. PMID 31180194
- [Result] Malvandi AM, Loretelli C, Ben Nasr M, Zuccotti GV, Fiorina P. Sitagliptin favorably modulates immune-relevant pathways in human beta cells. Pharmacol Res. 2019 Oct;148:104405. doi: 10.1016/j.phrs.2019.104405. Epub 2019 Aug 20. PMID 31442575
- [Result] Hu X, Liu S, Liu X, Zhang J, Liang Y, Li Y. DPP-4 (CD26) inhibitor sitagliptin exerts anti-inflammatory effects on rat insulinoma (RINm) cells via suppressing NF-kappaB activation. Endocrine. 2017 Mar;55(3):754-763. doi: 10.1007/s12020-016-1073-8. Epub 2016 Sep 9. PMID 27612849
- [Result] Ujhelyi J, Ujhelyi Z, Szalai A, Laszlo JF, Cayasso M, Vecsernyes M, Porszasz R. Analgesic and anti-inflammatory effectiveness of sitagliptin and vildagliptin in mice. Regul Pept. 2014 Nov;194-195:23-9. doi: 10.1016/j.regpep.2014.09.006. Epub 2014 Sep 16. PMID 25229125
- [Result] Matteucci E, Giampietro O. Dipeptidyl peptidase-4 (CD26): knowing the function before inhibiting the enzyme. Curr Med Chem. 2009;16(23):2943-51. doi: 10.2174/092986709788803114. PMID 19689275
- [Result] Jelsing J, Vrang N, van Witteloostuijn SB, Mark M, Klein T. The DPP4 inhibitor linagliptin delays the onset of diabetes and preserves beta-cell mass in non-obese diabetic mice. J Endocrinol. 2012 Sep;214(3):381-7. doi: 10.1530/JOE-11-0479. Epub 2012 Jul 3. PMID 22761275
- [Result] Kim SJ, Nian C, Doudet DJ, McIntosh CH. Dipeptidyl peptidase IV inhibition with MK0431 improves islet graft survival in diabetic NOD mice partially via T-cell modulation. Diabetes. 2009 Mar;58(3):641-51. doi: 10.2337/db08-1101. Epub 2008 Dec 10. PMID 19073764
- [Result] Davanso MR, Caliari-Oliveira C, Couri CEB, Covas DT, de Oliveira Leal AM, Voltarelli JC, Malmegrim KCR, Yaochite JNU. DPP-4 Inhibition Leads to Decreased Pancreatic Inflammatory Profile and Increased Frequency of Regulatory T Cells in Experimental Type 1 Diabetes. Inflammation. 2019 Apr;42(2):449-462. doi: 10.1007/s10753-018-00954-3. PMID 30707388
- [Result] Zhao Y, Yang L, Xiang Y, Liu L, Huang G, Long Z, Li X, Leslie RD, Wang X, Zhou Z. Dipeptidyl peptidase 4 inhibitor sitagliptin maintains beta-cell function in patients with recent-onset latent autoimmune diabetes in adults: one year prospective study. J Clin Endocrinol Metab. 2014 May;99(5):E876-80. doi: 10.1210/jc.2013-3633. Epub 2014 Jan 16. PMID 24432999
- [Result] Awata T, Shimada A, Maruyama T, Oikawa Y, Yasukawa N, Kurihara S, Miyashita Y, Hatano M, Ikegami Y, Matsuda M, Niwa M, Kazama Y, Tanaka S, Kobayashi T. Possible Long-Term Efficacy of Sitagliptin, a Dipeptidyl Peptidase-4 Inhibitor, for Slowly Progressive Type 1 Diabetes (SPIDDM) in the Stage of Non-Insulin-Dependency: An Open-Label Randomized Controlled Pilot Trial (SPAN-S). Diabetes Ther. 2017 Oct;8(5):1123-1134. doi: 10.1007/s13300-017-0299-7. Epub 2017 Sep 19. PMID 28929327
- See also: Related Info — https://www.niddk.nih.gov/about-niddk/strategic-plans-reports/diabetes-in-america-2nd-edition